CLINICAL TRIAL: NCT03833414
Title: Surgical Approach for Distal Humerus Fracture
Brief Title: Does Surgical-approach Affect Outcome After Fixation of Intra-articular Fractures of Distal Humerus?
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Aziz Hayder, admin assistant, Aga Khan University
Other Study IDs: 3799-Sur-ERC-15
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Distal Humerus Fracture
Keywords: intra-articular fractures; distal humerus; osteotomy; elbow joint
MeSH Terms: conditions — Humeral Fractures, Distal; Intra-Articular Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- (Group1): Triceps lifting approach .
  Interventions: Procedure: triceps lifting and olecranon osteotomy approaches
- (Group 2): olecranon osteotomy approach
  Interventions: Procedure: triceps lifting and olecranon osteotomy approaches

INTERVENTIONS:
Procedure: triceps lifting and olecranon osteotomy approaches — two different surgical approaches for distal humerus fracture

SUMMARY:
observational study at tertiary care hospital and level 1 trauma centre aiming to evaluate the difference between two common surgical approaches to distal humerus fracture fixation.

DETAILED DESCRIPTION:
Fractures around the distal humerus fractures make up to 2% of all fractures. Complex intra-articular distal humerus fractures present as challenge to restore of painless, stable and mobile elbow joint. Surgical exposure to all critical structures is of paramount importance to achieve anatomic reduction. Conflict still persists regarding the choice of ideal approach between triceps-sparing approach compared with olecranon osteotomy approach. In this study investigators compare the effect of surgical approach triceps lifting vs olecranon osteotomy on the functional outcome after fixation of distal humerus intra-articular fractures. Investigators conducted a non-funded, non-commercial, retrospective cohort study on participants with closed distal humerus intra-articular fractures between 2010 and 2015 at our tertiary care level-1 trauma and university hospital. Participants >18 years of age with closed complex intra-articular distal humerus fracture were operated using two different surgical approaches, either triceps lifting approach (Group1) or with olecranon osteotomy (Group 2). Functional evaluation of the participant is carried out with quick DASH scores at the final 1 year follow-up. Investigators concluded that triceps lifting approach can be used equally efficiently for exposure of these complex distal humerus injuries with no comprise in visibility of articular fragments.

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years of age with closed complex intra-articular distal humerus fracture (Intercondylar Fracture Riseborough Radin Classification type lll and lV) were included.

Exclusion Criteria:

* Patients with CVA (Cerebero-Vascular Accident), dementia and associated with neurovascular injuries which may impede with rehabilitation are excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all adult patients males and females who met the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Functional outcome using Quick DASH Score | 1 years followup
  Disabilities of Arm, Shoulder & Hand

IPD SHARING:
Plan to Share IPD: No
not allowed according to hospital policy